CLINICAL TRIAL: NCT01208844
Title: Cardiovascular Risk in Relation to Posttraumatic Stress Disorder in Young Women
Brief Title: Study of Physical Health for Women With Posttraumatic Stress or Depression
Status: Completed | Type: Observational
Sponsor: Nova Southeastern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeffrey Kibler, Ph.D., Professor, Nova Southeastern University
Other Study IDs: CPS06230812Exp.; 1R15HL085121-01A2 (NIH)
Record Dates: First submitted 2010-08-30; First posted 2010-09-24 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Healthy; Stress, Psychological; Depression; Posttraumatic Stress Disorders
MeSH Terms: conditions — Stress, Psychological; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Posttraumatic Stress
- Depression
- Healthy

SUMMARY:
The purpose of this study is to obtain a better understanding of how stress is related to health risks.

DETAILED DESCRIPTION:
Participants complete up to two study visits of approximately 3-4 hours each. The first study visit involves an interview about life experiences and emotions. If the participant is eligible for the second assessment, the average length of time between visit 1 and visit 2 will be 1-7 days. The second visit included physical measurements such as cholesterol and blood pressure, performing math and speaking tasks, and surveys to help us learn about healthy behaviors and emotions. No further follow-up of participants is conducted beyond the two study visits.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal
* Must be able to speak and read English fluently

Exclusion Criteria:

* Specific medications and chronic diseases
* History of heart attack (myocardial infarction)
* Pregnant or given birth in last 3 months
* Peri-menopausal or post-menopausal

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample, psychology clinics
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2008-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Number of Cardiovascular Risk Factors | Single assessment timepoint
  This primary outcome will be assessed at the second study visit (1-7 days from first study visit for those who are eligible).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Kibler, PhD, Principal Investigator — Nova Southeastern University
Locations (1):
- Center for Psychological Studies, Nova Southeastern University, Fort Lauderdale, Florida, United States